CLINICAL TRIAL: NCT04960982
Title: Changes in Testosterone, SHBG, DHEA and Cervical Length During Pregnancy in Egyptian Women With History of Recurrent Miscarriage
Brief Title: Changes in Pregnancy in Egyptian Women With History of Recurrent Miscarriage
Status: Completed | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Collaborators: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Essam El Mahdi, Dr, Kafrelsheikh University
Other Study IDs: 'RMPCOS2021
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS Recurrent Miscarriage
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PCOS-RM: PCOS women with history of RM
  Interventions: Diagnostic Test: blood test
- Non PCOS RM: Non PCOS women with history of RM
  Interventions: Diagnostic Test: blood test
- Control: women with no history of RM
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — blood sample is taken in first, second and third trimester of pregnancy

SUMMARY:
Introduction: Elevated levels of androgen and insulin-resistant have been implicated in recurrent miscarriage in women with PCOS. Published data are scarce on androgen level and cervical length of women with and without PCOS and a history of miscarriage.

Aim: The aim of this study was to investigate the levels of testosterone (TT), Sex Hormone Binding Globulin (SHBG), Dehyroepiandrostenedione (DHEA) and cervical length in Egyptian women with and without history PCOS and history of RM during pregnancy .

Method: Pregnant women with (n=38) and without (n=40) PCOS and history of recurrent miscarriages were recruited from the Obstetrics Department, Alagoza Hospital, Cairo, Egypt. Healthy pregnant women without PCOS and history of RM (n=40, HC) were also recruited. TT, SHBG,DHEA and Sex Hormone Binding Globulin (SHBG) level and cervical length were assessed at first, second and the third trimester or at the start of miscarriage

DETAILED DESCRIPTION:
Introduction

Recurrent miscarriage (RM )is defined as the loss of three of more consecutive pregnancies before 20 weeks gestation (Royal College of Obstetricians & Gynaecologists 2011, Practice Committee of American Society for Reproductive Medicine 2013). The prevalence of RM varies from country to country and within communities within the country. It tends to be higher in developing countries. However it effects 1% to 2%of women (Jeve et al., 2014, Green-top Guideline No. 17).Other studies have reported incidences of RM between 0.5% and 2.3 % (Christiansen et al.,2007, Stirrat et al., 1990, Alberman et al., 1988).

Currently the established risk factors of RM include hormonal associated conditions (Stephenson et al.,1996, Fox-Lee et al., 2007) , uterine abnormalities (including adhesions post-surgery) (Rimbizis et al.,2001, Salim et al.,2003) anti-phospholipid syndrome Thrombotic (Greer et al., 2003) , chromosomal and genetic (Braekeleer et al., 1990 , Clifford et al.,1994, Stephenson et al., 2006, Franssen et al., 2006) conditions .Indeed some researchers consider PCOS as a risk factor, However some don't.

Approximately 8% to 12% of RM is due to endocrine causes mainly due to hyperandrogenism and hyperinsulinemia in PCOS (Smith et al., 2011, Witchel et al., 2019, Rai et al., 2000) . Little research focuses directly on the effect of PCOS during gestation and how that can be linked to poor pregnancy outcomes. However, there is a positive correlation between increased risk of miscarriage and hyperhomocysteinemia in insulin resistant patients, a common component of PCOS (Chakraborty et al.,2013).

The current literature providing conflicting views on androgen levels effecting pregnancy in PCOS patients some clarity is required as to whether its elevation impacts pregnancy. Not only that, but the is limited published data which compared the androgen and cervical length at different gestational periods of women with history of miscarriage either due to PCOS or for unknown reasons.

Cervical cerclage (CC) is one of the management options offered to patient who has history of midterm miscarriage. The efficacy of CC in management is still doubtable.

Aim The aim of this study was to investigate the levels of testosterone (TT), Sex Hormone Binding Globulin (SHBG), Dehyroepiandrostenedione (DHEA) and cervical length in women with and without history PCOS and history of RM during pregnancy .

Subjects and Methods

- Subjects

Participants of the study are women with (n=38) and without PCOS (n=40) and history of RM were recruited during their first antenatal visit from Al-Agoza Hospital, Cairo, Egypt. They were recruited during their first antenatal visit. Similarly pregnant women without PCOS (n=40) with no history of RM were recruited. Detailed demographic, medical and obstetric history was documented.

The inclusion criteria for the study were women aged 23 to 40 years at the time of enrolment into the study. The exclusion criteria for all participants included any other diagnosed medical condition link with increased risk of miscarriage, including thyroid status and gestational diabetes. All participants examined at the time of recruitment.

The control group were matched for age and BMI with no previous history of RM.

This study was conducted in line with the human experimentation guidelines, dictated by the Helsinki declaration. The procedures used were approved by local ethical committee and conducted in line with the practices of Al-Agoza Hospital, Cairo, Egypt. All patients within the study were briefed on the procedures and protocol that would take place and written consent was obtained before induction into the study.

- Methods

Confirmation of the pregnancy was made by beta-human chorionic gonadotrophin (Bhcg ) plus ultrasound scan and clinical history in case of miscarriage.

Diagnosis for patients with recurrent miscarriage was in concordance with the guidelines defined by the Royal College of Obstetricians and Gynaecologists; the loss of three or more consecutive pregnancies (Royal College of Obstetricians & Gynaecologists 2011 ).The diagnosis of PCOS was based on Rotterdam 2003 Criteria (Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group 2004 ) which require two of the following; Oligo- or anovulation, Clinical and/or biochemical signs of hyperandrogenism or Polycystic ovaries and exclusion of other related disorders.

Blood Samples were collected by a professional trained in phlebotomy at the time points ; first, second and the third trimester or at the start of miscarriage .Samples were analysed for TT, SHBG,SHBG and DHEA using The ADVIA Centaur® XPT Immunoassay System - Siemens (https://www.siemens-healthineers.com/en-uk/immunoassay/systems/advia-centaur-xpt#TECHNICAL_SPECIFICATIONS).This system is easy to use where samples and reagents which could be loaded or without pausing the system. Also it doesn't require daily set up procedure and implement new assays immediately with one easy scan of a test definition bar code.

It requires 10-200 μL per test. it offers Automatic dilution varies by assay, up to 1:2500. The reagent capacity on board is 30 assays.

Similarly, cervical length was also measured at first, second and the third trimester or at the start of miscarriage .It was measured via transvaginal ultrasound (Berghella et al.,1997). The Voluson™ E8 ultrasound system is used for this study (https://www.gehealthcare.com/products/ultrasound/voluson/voluson-e8 ). The data was recorded by measuring the distance between the external os of the cervix and to where the cervix is closed defined by the apex of the funnelling of the membranes (Berghella et al., 1997) .

All patients within the RM groups attended cerclage treatment during the second trimester, this included elective and emergency elective procedures. Patients presented at the time of delivery or for recording of miscarriage where gestational age, gender of the fetus/baby and whether it was a live birth was noted.

ELIGIBILITY:
Inclusion Criteria: women aged 23 to 40 years at the time of enrolment into the study. The exclusion criteria for all participants included

Exclusion Criteria:

Any other diagnosed medical condition link with increased risk of miscarriage, including thyroid status and gestational diabetes

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Egyptian women
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Cervical length changes during pregnancy | 9 months
  Cervical length is shorter in recurrent miscarriage groups at the start of the study and getting shorter during pregnancy
Androgens changes during pregnancy | 9 months
  TT, SHBG,DHEA and Sex Hormone Binding Globulin (SHBG) level were assessed at first, second and the third trimester or at the start of miscarriage

CONTACTS AND LOCATIONS:
Overall Officials: Essam El Mahdi, MD, Principal Investigator — London Metropolitan University
Locations (1):
- Kafrelsheikh University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
when study complited we will decide